CLINICAL TRIAL: NCT05705375
Title: Understanding the Effect of Waterpipe Size on Smoking Behavior, Toxicant Exposures and Subjective Experiences
Brief Title: Effect of Waterpipe Size on Smoking Behavior and Exposures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0458
Record Dates: First submitted 2022-12-22; First posted 2023-01-30 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-09

CONDITIONS: Waterpipe Size

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- waterpipe regular smokers (Experimental): waterpipe regular smokers will be invited for 3 lab visits where they are allocated (random order) to smoke 3 waterpipe different sizes.
  Interventions: Other: Waterpipe size

INTERVENTIONS:
Other: Waterpipe size — Participants will have 3 lab visits where they are allocated (random order) to smoke a small waterpipe in one visit, smoke a medium waterpipe in a second visit and smoke a large waterpipe in a third visit.

SUMMARY:
The goal of this clinical trial is to learn how waterpipe (WP) size affects smoking behavior, toxicant exposure, and subjective experiences in young adult WP smokers (ages 21-39). The main questions it aims to answer are:

* Does WP size change puffing behavior?
* Does WP size change exposure to nicotine and carbon monoxide?
* Does WP size change perceptions of harm, satisfaction, craving, or withdrawal?

Participants will smoke small, medium, and large WPs in separate sessions. Researchers will measure puffing behavior, saliva nicotine, exhaled carbon monoxide, and survey responses before and after each session.

DETAILED DESCRIPTION:
This study will examine the effect of waterpipe (WP) size manipulation on smoking behavior, toxicant exposure, and subjective experiences among young adult WP smokers. A total of 40 participants ages 21-39 will complete a 2x3 crossover design, where the within-subject factors are time (pre vs. post WP smoking) and study condition (small vs. medium vs. large). Each participant will attend three 45-minute laboratory sessions, each using a different WP size.

Aim 1: To examine the effect of WP size on puffing behavior and toxicant exposure. Puff topography parameters (puff number, duration, average puff volume, total inhaled volume, and inter-puff interval) will be measured during smoking. Exhaled CO and saliva nicotine concentrations will be measured pre- and post-session.

Aim 2: To examine the effect of WP size on harm perception and subjective experiences. Outcomes include harm perception, WP Evaluation Scale, Duke Sensory Questionnaire, Questionnaire of Smoking Urges (brief), and Minnesota Nicotine Withdrawal Scale.

This project will generate novel evidence on how WP size influences smoking behavior, exposure to nicotine and CO, and user perceptions. Findings will inform the FDA on the potential impact of WP size regulation and help guide the development of size-specific standards to protect public health.

ELIGIBILITY:
Inclusion Criteria:

* regular waterpipe smokers (smoking at least once a week for the past 6 months)
* generally healthy and
* able to provide written informed consent; and willing to attend the 3 lab sessions

Exclusion Criteria:

* history of chronic diseases such as diabetes, high blood cholesterol, hepatic disease
* respiratory chronic diseases
* cardiovascular diseases including low or high blood pressure (BP)

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Small → Medium → Large: Participants first smoke the small WP in Session 1, followed by the medium WP in Session 2, and the large WP in Session 3. Each session lasts 45 minutes and is separated by a 48-hour washout period.
- Small → Large → Medium: Participants first smoke the small WP, then the large WP, and finally the medium WP, with each 45-minute session separated by a 48-hour washout.
- Medium → Large → Small: Participants first smoke the medium WP, then the large WP, and finally the small WP, with each 45-minute session separated by a 48-hour washout.
- Medium → Small → Large: Participants first smoke the medium WP, then the small WP, and finally the large WP, with each 45-minute session separated by a 48-hour washout.
- Large → Medium → Small: Participants first smoke the large WP, then the medium WP, and finally the small WP, with each 45-minute session separated by a 48-hour washout.
- Large → Small → Medium: Participants first smoke the large WP, then the small WP, and finally the medium WP, with each 45-minute session separated by a 48-hour washout.
Period: First Intervention (1 Day)
Arm/Group | Small → Medium → Large | Small → Large → Medium | Medium → Large → Small | Medium → Small → Large | Large → Medium → Small | Large → Small → Medium
Started | 3 | 7 | 11 | 6 | 6 | 7
Completed | 3 | 7 | 11 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (48 Hours)
Arm/Group | Small → Medium → Large | Small → Large → Medium | Medium → Large → Small | Medium → Small → Large | Large → Medium → Small | Large → Small → Medium
Started | 3 | 7 | 11 | 6 | 6 | 7
Completed | 3 | 7 | 11 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Small → Medium → Large | Small → Large → Medium | Medium → Large → Small | Medium → Small → Large | Large → Medium → Small | Large → Small → Medium
Started | 3 | 7 | 11 | 6 | 6 | 7
Completed | 3 | 7 | 11 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (48 Hours)
Arm/Group | Small → Medium → Large | Small → Large → Medium | Medium → Large → Small | Medium → Small → Large | Large → Medium → Small | Large → Small → Medium
Started | 3 | 7 | 11 | 6 | 6 | 7
Completed | 3 | 7 | 11 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Small → Medium → Large | Small → Large → Medium | Medium → Large → Small | Medium → Small → Large | Large → Medium → Small | Large → Small → Medium
Started | 3 | 7 | 11 | 6 | 6 | 7
Completed | 3 | 7 | 11 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: waterpipe regular smokers will be invited for 3 lab visits where they are allocated (random order) to smoke 3 waterpipe different sizes.
Arm/Group | Waterpipe Regular Smokers
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Saliva Nicotine [Mean (Standard Deviation); unit: ng/mL] | 9 (3.5)
Exhaled Carbon Monoxide [Mean (Standard Deviation); unit: PPM] | 1.2 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Waterpipe Evaluation Scale
Description: An 11-item questionnaire assessing participants' subjective experience of smoking waterpipe (WP) tobacco. Each item is scored on a 7-point Likert scale (1 = "not at all" to 7 = "extremely"). For analysis, item scores were averaged across the 11 items to produce a mean WES score for each WP size, with higher scores indicating a more satisfactory smoking experience. The scale captures aspects such as satisfaction, taste, cravings, and sensory enjoyment in the throat and chest.
Time Frame: Immediately after the exposure (smoking)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Small Waterpipe; Medium Waterpipe; Large Waterpipe: waterpipe regular smokers attended 3 lab visits where they are allocated (random order) to smoke 3 waterpipe different sizes.
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 4.2 (0.8) | 4.4 (0.7) | 4.7 (0.8)

2. Primary Outcome: Duke Sensory Questionnaire
Description: A 9-item questionnaire assessing participants' sensory experience of smoking waterpipe (WP) tobacco. Each item is scored on a 7-point Likert scale (1 = "not at all" to 7 = "extremely"). Item scores were averaged across the 9 items to produce a mean DSQ score for each WP size, with higher scores indicating a more positive sensory experience (e.g., satisfaction, perceived nicotine strength, and puff intensity).
Time Frame: Immediately after the exposure (smoking)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 4.4 (0.9) | 4.0 (0.8) | 3.8 (0.9)

3. Primary Outcome: Harm Perception Questionnaire
Description: This is a 3-item scale assessing participants' perception of the harmfulness of waterpipe (WP) tobacco smoking. Each item is scored on a 7-point Likert scale ranging from 1 = "a lot less harmful" to 7 = "a lot more harmful." Item scores were averaged across the 3 items to produce a mean harm perception score for each WP size, with higher scores indicating greater perceived harm.
Time Frame: Immediately after the exposure (smoking)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 3.5 (0.5) | 3.7 (0.2) | 3.8 (0.2)

4. Primary Outcome: Saliva Nicotine
Description: How participants' nicotine concentrations change based on the different smoked waterpipe sizes
Time Frame: Immediately after the exposure (smoking)
Population: A small number of participants could not provide adequate saliva nicotine samples due to technical issues encountered during the collection process
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 36 | 36 | 36
ng/mL | 1065.5 (247.4) | 620.2 (123.2) | 701.4 (118.9)

5. Primary Outcome: Puff Topography: Smoking Time
Description: The total time spent smoking during a single WP session, measured in minutes. Longer times indicate greater duration of smoking across WP sizes.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
Minutes | 38.05 (5.82) | 35.5 (7.23) | 36.27 (7.23)

6. Primary Outcome: Puff Topography: Cumulative Puff Time
Description: The total time spent actively inhaling smoke across all puffs in a WP session, measured in minutes using a puff topography device. Higher values indicate more total inhalation time.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
Minutes | 5.10 (2.67) | 5.10 (2.95) | 6.67 (4.02)

7. Primary Outcome: Puff Topography: Puff Duration
Description: The average length of each puff in seconds, measured using a puff topography device in the WP hose. Longer puff duration indicates deeper inhalation per puff.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
Seconds | 2.15 (1.08) | 2.20 (1.03) | 2.45 (0.96)

8. Primary Outcome: Puff Topography: Average Flow Rate
Description: The average rate of smoke inhaled per second during puffing, measured in liters per minute with a puff topography device. Higher flow rates indicate faster inhalation.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
L/min | 15.14 (6.11) | 16.65 (6.05) | 18.92 (7.96)

9. Primary Outcome: Puff Topography: Number of Puffs
Description: The total number of puffs taken during a WP session, measured using a puff topography device. Higher counts indicate more frequent puffing.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: Puffs
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
Puffs | 161.05 (90.39) | 162.31 (122.51) | 182.90 (138.46)

10. Primary Outcome: Puff Topography: Total Smoke Volume Inhaled
Description: Total smoke inhaled during a single WP session, measured in liters using a puff topography device in the WP hose. Higher values indicate greater smoke intake across WP sizes.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
Liters | 76.82 (50.67) | 79.85 (48.27) | 116.19 (63.18)

11. Primary Outcome: Puff Topography: Puff Volume Average
Description: Mean volume of each puff during a WP session, measured in liters using a puff topography device in the WP hose. Higher values indicate larger puff sizes across WP sizes.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
Liters | 0.57 (0.39) | 0.64 (0.45) | 0.78 (0.42)

12. Primary Outcome: Puff Topography: Maximum Puff Volume
Description: The largest single puff volume inhaled during a WP session, measured in liters using a puff topography device. Higher values indicate the strongest inhalation effort across puffs.
Time Frame: During the exposure (smoking), up to 45 mins
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
Number analyzed (Participants) | 40 | 40 | 40
Liters | 1.21 (0.50) | 1.34 (0.64) | 1.62 (0.62)

ADVERSE EVENTS:
Time Frame: Each participant was monitored during and immediately after three laboratory smoking sessions (~45 minutes each) separated by ≥48 hours (~1 week total monitoring per participant). This monitoring process was carried out for all participants over the approximate 23-month study period.
Arm/Group | Small Waterpipe | Medium Waterpipe | Large Waterpipe
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT05705375/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT05705375/ICF_000.pdf